CLINICAL TRIAL: NCT04287283
Title: The Profile of Cognitive Function of Patients Who Had Neurocognitive Evaluation at the Sagol Center for Hyperbaric Medicine and Research
Brief Title: Cognitive Profile of Patients at the Sagol Center for Hyperbaric Medicine and Research
Status: Active, not recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shay Efrati, Prof., Assaf-Harofeh Medical Center
Other Study IDs: ASF-19-0267
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: TBI (Traumatic Brain Injury); Stroke; Fibromyalgia; Aging
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke; Fibromyalgia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBOT: Patients with chronic brain injury or cognitive complaints that have been treated with Hyperbaric oxygen therapy and underwent computerized cognitive tests before and after the treatment
  Interventions: Other: Hyperbaric Oxygen

INTERVENTIONS:
Other: Hyperbaric Oxygen — 40-60 daily hyperbaric sessions, 5 days per week. Each session consists of 90 minutes exposure to 100% oxygen at 1.5-2 ATA.

SUMMARY:
In the investigator's institute there is ongoing treatment of different patients with cognitive deficits using Hyperbaric oxygen therapy (HBOT). These patients undergo neuro-cognitive function computerized tests before and after treatment.

The aim of this study was to retrospectively evaluate the cognitive changes before and after HBOT in different patients populations.

DETAILED DESCRIPTION:
Retrospective analysis of patients suffering from chronic neuro-cognitive deficits due to different conditions, treated at Sagol center for hyperbaric medicine and research, Shamir (Assaf Harofeh) Medical Center, Israel

Patients included if they had at least two neurocognitive tests, before and after Hyperbaric Oxygen Therapy (HBOT). The study was approved by the institutional review board of the hospital.

Patients were treated with 40-60 daily hyperbaric sessions, 5 days per week. Each session consists of 90 minutes exposure to 100% oxygen at 1.5-2 ATA.

ELIGIBILITY:
Inclusion Criteria:

* Patients included if they completed at least two neuro-cognitive computerized tests, before and after HBOT

Exclusion Criteria:

* Patients who were not able to complete two cognitive tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective analysis of patients suffering from chronic neuro-cognitive damage or complaints treated at Sagol center for hyperbaric medicine and research, Shamir (Assaf Harofeh) Medical Center, Israel since 2008 .
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive scores | baseline and 12 weeks
  change in scores in a computerized neuro-cognitive test, "IQ-scale" score, normalized for age and education, with mean=100 and SD=15 points in healthy population, higher score implies better results.

CONTACTS AND LOCATIONS:
Locations (1):
- hyperbaric center Asaf harofe medical center, Rishon LeZiyyon, Israel

IPD SHARING:
Plan to Share IPD: Undecided